CLINICAL TRIAL: NCT06035276
Title: Sample Collection for Biosensor Development Using Real-world Conditions With Exposure to "Urban" Versus "Clean" Air in Healthy Subjects and COPD Patients.
Brief Title: Biosensor and Environmental Sensor Development Within the REMEDIA Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23-01 REMEDIA-2
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Healthy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This study is a single-center research project with a 2-period, sequential, cross-over ("clean" vs. versus "urban" air) design, which supports the development of the REMEDIA sensor toolkit with clinically relevant data and bio samples. The approach is exploratory, blinding or randomization are not applicable. Two populations will participate: healthy subjects and COPD subjects with GOLD stage 1 to 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy subjects (Other)
  Interventions: Other: Exposure to clean air; Other: Exposure to urban air
- COPD patients (Other)
  Interventions: Other: Exposure to clean air; Other: Exposure to urban air

INTERVENTIONS:
Other: Exposure to clean air — Subjects will be exposed to filtered indoor air ("clean" air) for 4 hours in the Fraunhofer Environmental Exposure Chamber. The chamber can accommodate up to 18 subjects, is ventilated by HEPA-filtered and conditioned air, ensuring a constant humidity (40 ± 10%), temperature (22 ± 2°C), and airflow (1500 ± 100 m3/hr). During exposure they will perform an intermittent bicycle ergometer activity at 50 W for 10 minutes alternating with 20 minutes rest.
Other: Exposure to urban air — Subjects will be brought to a traffic dense urban region ("urban air") with high traffic density and increased levels of particulate matter and vehicle emissions. Subjects will stay in this area for 4 hours. During exposure, all subjects will walk together with study staff. Rest periods are only allowed outside. Intervals of activity and rest will be similar to the "clean air" regimen.

SUMMARY:
The aim of this proof-of-concept study is to obtain data that will contribute to the development of sensor devices (biosensor and environmental sensor) for patients with lung diseases (e.g. COPD). The study aims to validate our previous results from healthy subjects by joint testing of the biosensor and environmental device in a real-world setting. Healthy subjects and COPD subjects will be exposed to air of a traffic dense urban region ("urban" air) and to filtered indoor air ("clean" air) during activity and rest. Environmental and biomarker sensors will be used to measure several biomarkers and environmental conditions.

DETAILED DESCRIPTION:
The EU-sponsored REMEDIA project (Impact of exposome on the course of lung diseases, Grant agreement ID 874753) contributes to the understanding of the influence of the exposome on chronic obstructive pulmonary disease (COPD) and cystic fibrosis (CF). While COPD is considered to be mainly related to the external exposome (smoking, ambient particulate matter, household air pollution, occupational particulate matter, ozone and second-hand smoke) CF is the consequence of a genetic defect in the CFTR gene, which gives an essential role to factors outside of the exposome. However, COPD and CF share common characteristics such as high phenotypic variability of unknown origin, and similar progressive loss of lung function with small bronchi alterations. Given this high phenotypic variability it is clear that the overall picture must be supplemented by considering additional components of the exposome. The REMEDIA project investigates the specific exposome associated with particular COPD or CF phenotypes.

Objective of work package 3 within the REMEDIA project is the development of a mobile environmental sensor toolbox that is capable to assess the external exposome (temperature, humidity, particulate matter (PM), volatile organic compounds (VOC), nitrogen dioxide (NO2), ozone (O3), carbon-monoxide (CO), and sulfur dioxide (SO2)) and a mobile biosensor unit that can measure inflammatory biomarkers in exhaled breath. Currently specific sensors for the analysis of hexanal, nitrotyrosine and neutrophils elastase are included into the sensor tool kit. Other relevant molecules are evaluated and selected in other work packages and could be included into the tool kit.

Our previous experimental exposure study focused on the major environmental air pollutant ozone and was supposed to test the biosensor unit under close to "real life conditions". Ozone is known to cause a temporary neutrophilic airway inflammation, which is also typical for patients with COPD and CF.

This proof-of-concept study aims to validate our previous results from healthy subjects by joint testing of the biosensor and environmental device in a real-world setting. Healthy subjects and COPD subjects will be exposed to air of a traffic dense urban region ("urban" air) and to filtered indoor air ("clean" air) during activity and rest. The biosensor will measure the following biomarker: 3-Nitrotyrosin, Hexanal and Neutrophil Elastase. The environmental sensor will measure the following parameters: CO, O3, SO2, NO2, VOC, PM10, PM2.5, temperature, humidity, light and sound level. The collected data will be evaluated in terms of population and exposure.

ELIGIBILITY:
Inclusion criteria:

Healthy subjects:

1. Able and willing to give written informed consent.
2. Healthy male and female subjects aged 40-70 years, inclusive. Women will be considered for inclusion if they are:

   Not pregnant, as confirmed by pregnancy test (see assessment schedule), and not breastfeeding.

   Of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is postmenopausal, with documented proof of hysterectomy or tubal ligation, without an alternative medical cause according to the Clinical Trial Facilitation Group (CTFG) document "Recommendations related to contraception and pregnancy testing in clinical trials").

   Of childbearing potential and using a highly effective method of contraception according to the contraception requirements in section 7.2 from two weeks prior to visit 1 until the end of study participation.
3. Normal lung function with FEV1 predicted ≥ 80% and FEV1/FVC≥70%.
4. Body mass index of ≥18.6 and ≤30 kg/m2
5. Non-smoker or former smoker with <10 pack years who had stopped smoking (including e-cigarettes) for at least 12 months before Screening.

COPD subjects:

1. Able and willing to give written informed consent.
2. Male and female subjects aged 40-70 years, inclusive. Women will be considered for inclusion if they are:

   Not pregnant, as confirmed by pregnancy test (see assessment schedule), and not breastfeeding.

   Of non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is postmenopausal, with documented proof of hysterectomy or tubal ligation, without an alternative medical cause according to the Clinical Trial Facilitation Group (CTFG) document "Recommendations related to contraception and pregnancy testing in clinical trials").

   Of childbearing potential and using a highly effective method of contraception according to the contraception requirements in section 7.2 from two weeks prior to visit 1 until the end of study participation.
3. Clinical diagnosis of COPD stage 1 to 2 (GOLD classification)
4. FEV1/FVC <70% post-bronchodilator at visit 1
5. FEV1 ≥50% of the predicted normal value post-bronchodilator at visit 1
6. FEV1 ≥1.5L pre-bronchodilator
7. Ex-smokers for at least 12 months with a history of at least 10 pack years.
8. Body mass index of ≥ 18.6 and ≤30 kg/m2.

Exclusion criteria:

Healthy subjects:

1. Past or present disease, which as judged by the investigator, may affect the outcome of the study or put the subject at risk because of participation in the study. These diseases include, but are not limited to, coagulation disorders, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis)
2. Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for short term pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements.
3. Clinically relevant allergy against airborne allergens (such as pollen).
4. Infections of the lower respiratory tract within 4 weeks prior to screening
5. Infections of the upper respiratory tract within 2 weeks prior to screening
6. Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, lung function, or ECG at Visit 1, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study.
7. Positive drug screen for methadone, cannabis, opiates, cocaine metabolites, amphetamines, barbiturates and benzodiazepines at visit 1
8. History of drug or alcohol abuse
9. Risk of non-compliance with study procedures
10. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study

COPD subjects:

1. Past or present disease other than COPD, which as judged by the investigator, may affect the outcome of the study or put the subject at risk because of participation in the study. These diseases include, but are not limited to, coagulation disorders cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis).
2. Regular intake of any prescribed or over the counter medication, which as judged by the investigator, may affect the outcome of the study or put the subject at risk because of participation in the study. Explicitly not allowed is treatment with GCS, NSAIDs or any other anti-inflammatory medication. Explicitly allowed is treatment with SABA/LABA/LAMA, paracetamol for pain relief, antihypertensives, lipid-lowering medications, antidiabetics, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements.
3. Clinically relevant allergy against airborne allergens (such as pollen).
4. Infections of the lower respiratory tract within 4 weeks prior to screening.
5. Infections of the upper respiratory tract within 2 weeks prior to screening
6. Exacerbation of COPD (treatment with oral or parenteral antibiotics and/or oral or parenteral GCS and/or hospitalization related to COPD) within 60 days before visit 1.
7. Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, lung function, or ECG at visit 1, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study.
8. Positive drug screen for methadone, cannabis, opiates, cocaine metabolites, amphetamines, barbiturates and benzodiazepines at visit 1.
9. History of drug or alcohol abuse.
10. Risk of non-compliance with study procedures.
11. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Concentration of Biomarkers in exhaled breath condensate collected by biosensor | On day 1,3,5,8,10, and 12 of the study
  3-Nitrotyrosin
Concentration of Biomarkers in exhaled breath condensate collected by biosensor | On day 1,3,5,8,10, and 12 of the study
  Hexanal
Concentration of Biomarkers in exhaled breath condensate collected by biosensor | On day 1,3,5,8,10, and 12 of the study
  Neutrophil Elastase
Data collected by environmental sensor | Through study completion (study days 1-12)
  Concentration of CO
Data collected by environmental sensor | Through study completion (study days 1-12)
  Concentration of O3
Data collected by environmental sensor | Through study completion (study days 1-12)
  Concentration of SO2
Data collected by environmental sensor | Through study completion (study days 1-12)
  Concentration of NO2
Data collected by environmental sensor | Through study completion (study days 1-12)
  Concentration of VOC
Data collected by environmental sensor | Through study completion (study days 1-12)
  Concentration of PM10
Data collected by environmental sensor | Through study completion (study days 1-12)
  Concentration of PM2.5
Data collected by environmental sensor | Through study completion (study days 1-12)
  temperature
Data collected by environmental sensor | Through study completion (study days 1-12)
  Humidity of the subject's ambient air within a range of 0 % to 100 % and with a resolution of 1 %
Data collected by environmental sensor | Through study completion (study days 1-12)
  Light level of the subject's environment within a range of 350 nm to 1100 nm
Data collected by environmental sensor | Through study completion (study days 1-12)
  Sound level of the subject's environment within a range of 20 Hz to 10 kHz and with a resolution of 1 Pa / 1 kHz

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez Fernandez E, De Santi C, De Rose V, Greene CM. CFTR dysfunction in cystic fibrosis and chronic obstructive pulmonary disease. Expert Rev Respir Med. 2018 Jun;12(6):483-492. doi: 10.1080/17476348.2018.1475235. Epub 2018 May 23. PMID 29750581
- [Background] De Rose V, Molloy K, Gohy S, Pilette C, Greene CM. Airway Epithelium Dysfunction in Cystic Fibrosis and COPD. Mediators Inflamm. 2018 Apr 8;2018:1309746. doi: 10.1155/2018/1309746. eCollection 2018. PMID 29849481
- [Background] Holz O, Jorres RA, Timm P, Mucke M, Richter K, Koschyk S, Magnussen H. Ozone-induced airway inflammatory changes differ between individuals and are reproducible. Am J Respir Crit Care Med. 1999 Mar;159(3):776-84. doi: 10.1164/ajrccm.159.3.9806098. PMID 10051250